CLINICAL TRIAL: NCT03760952
Title: Human Leukocyte Antigen Typing and Tumor Antigen Expression Profiling
Status: Completed | Type: Observational
Sponsor: Immatics US, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IMA-SCREENING
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Refractory Cancer; Recurrent Cancer; Adult Solid Tumor; Neoplasms
Keywords: T-cell therapy; Immunotherapy; Screening; Metastatic; Previously Treated
MeSH Terms: conditions — Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This screening study will identify HLA molecular subtype positive and tumor antigen target(s) positive patients who may be eligible for enrollment into Immatics clinical studies. This screening study is intended for patients with advanced and/or metastatic solid cancers. No treatment intervention will occur as part of this screening study.

DETAILED DESCRIPTION:
The purpose of this screening study is to identify human leukocyte antigen (HLA) molecular subtype positive and tumor antigen target(s) positive patients. No treatment intervention will occur as part of this screening study.

After diagnosis of advanced and/or solid metastatic cancers, patients will be tested for HLA molecular subtype positivity. Patients that are HLA molecular subtype positive are then assessed to determine if their tumor antigen target(s) is positive (biopsy screening). Fresh tumor tissue obtained by a biopsy for this screening study will be required. If the patient is undergoing a surgical procedure directed towards tumor or palliative treatment (e.g., a resection, debulking surgery, etc.) and has consented to the study, then fresh tissue may be collected during the procedure to avoid the patient being subjected to another biopsy.

Tumor antigen targets in fresh tumor samples will be determined by an in vitro diagnostic (IVD) assay. Therefore, any remaining tumor specimens may be used for exploratory biomarker analyses and validation studies for regulatory approval.

Immatics is conducting clinical studies which target patients with advanced and/or metastatic solid cancers. Patients who are HLA subtype phenotype positive and whose tumors express one or more of the tumor antigen targets of interest may be eligible for ongoing clinical studies of adoptive cell therapy (ACT).

ELIGIBILITY:
Inclusion Criteria:

1. Signed an Informed Consent Form (ICF)
2. Patients ≥ 18 years of age
3. Patients with confirmed advanced and/or metastatic solid tumors.
4. For liver cancer patients, the diagnosis must be confirmed

   * Pathological diagnosis of liver cancer based on biopsy/resection is required
   * For patients without pathological diagnosis, an imaging technique obtained by computed tomography (CT) scan or magnetic resonance imaging (MRI) is needed.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 0-1
6. Life expectancy > 6 months
7. There is no limitation for prior anti-cancer treatments
8. HLA molecular phenotype positive.
9. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST)1.1
10. At least one lesion considered accessible for biopsy unless fresh tumor tissue is being collected during a surgical procedure directed towards tumor treatment or palliative therapy or the patient has uterine cancer (including endometrial cancer or uterine carcinosarcoma) or melanoma
11. Patient has adequate pulmonary function
12. Acceptable organ and marrow function
13. Acceptable coagulation status
14. Adequate hepatic function
15. Acceptable levels of serum creatinine
16. For liver cancer patients only, Child-Pugh score of < 6

Exclusion Criteria:

1. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
2. Patients with primary central nervous system (CNS)/brain tumors
3. Patients whose tumors have very low expression of tumor antigen targets such as kidney chromophobe, thyroid carcinoma, and prostate adenocarcinoma
4. Patients who are pregnant or are breastfeeding
5. Patients with serious autoimmune disease Note: At the discretion of the investigator, these patients may be included if their disease is well controlled without the use of immunosuppressive agents
6. Patients with prior stem cell transplantation or solid organ transplantation
7. Any condition contraindicating leukapheresis
8. Patients with any of the following cardiac conditions: uncontrolled hypertension despite optimal therapy, uncontrolled angina, ventricular arrhythmias, congestive heart failure, baseline left ventricular ejection fraction ≤ 50%, prior or current cardiomyopathy, atrial fibrillation with heart rate > 100 bpm, unstable ischemic heart disease
9. Patients with active diverticulitis, intra-abdominal abscess, or GI obstruction
10. Patients with active pneumonitis
11. Patients with active (uncontrolled/untreated) brain metastases NOTE: Patients with a history of brain metastases may be eligible, if an imaging scan with contrast enhancement not older than 4 weeks is able to exclude the existence of currently active brain metastasis.
12. History of hypersensitivity on fludarabine (FLU), cyclophosphamide (CY), or interleukin (IL)-2
13. History of current immunodeficiency disease or prior treatment compromising immune function at the discretion of the investigator.
14. Patients with Grade 3 or Grade 4 immune-related toxicities related to checkpoint inhibitors or patients requiring corticosteroid treatment (≥ 10 mg/day prednisone or equivalent dose).
15. Patients with bleeding diathesis or coagulopathy
16. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with patient's safety
17. HIV infection, active hepatitis B or C infection. History of treated hepatitis B or C is permitted if the viral load is undetectable per qPCR and/or nucleic acid testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed advanced and/or metastatic solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with protocol-specified HLA subtype | 3 years
Frequency of patients with expression of analyzed tumor antigen targets | 3 years

OTHER OUTCOMES:
Incidence of antigen target expression in solid tumors | 3 years
Comparison of antigen target expression in fresh and FFPE tumor samples | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, M.D., Study Director — Immatics US
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Oncology Consultants, Houston, Texas